CLINICAL TRIAL: NCT03595618
Title: Efficacy and Safety of 3 Doses of S201086/GLPG1972 Administered Orally Once Daily in Patients With Knee Osteoarthritis. A 52-week International, Multi-regional, Multi-center, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study
Brief Title: A Study to Assess Efficacy and Safety of GLPG1972/S201086 in Participants With Knee Osteoarthritis
Acronym: Roccella
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Collaborators: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG1972-CL-201; 2017-004581-10 (EudraCT Number); U1111-1205-0321 (Other: Universal Trial Number)
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Results first posted 2021-05-12 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GLPG1972 75 mg (Experimental): Participants received 1 film-coated tablet of GLPG1972 75 mg and 3 GLPG1972 matching placebo tablets, orally once daily for 52 weeks.
  Interventions: Drug: GLPG1972; Drug: Placebo
- GLPG1972 150 mg (Experimental): Participants received 2 film-coated tablets of GLPG1972 75 mg (total dose 150 mg) and 2 GLPG1972 matching placebo tablets, orally once daily for 52 weeks.
  Interventions: Drug: GLPG1972; Drug: Placebo
- GLPG1972 300 mg (Experimental): Participants received 4 film-coated tablets of GLPG1972 75 mg (total dose 300 mg), orally once daily for 52 weeks.
  Interventions: Drug: GLPG1972
- Placebo (Placebo Comparator): Participants received 4 film-coated tablets of GLPG1972 matching placebo, orally once daily for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG1972 — Film-coated tablets of GLPG1972 for oral use.
  Arms: GLPG1972 150 mg; GLPG1972 300 mg; GLPG1972 75 mg
Drug: Placebo — Film-coated tablets of matching placebo for oral use.
  Arms: GLPG1972 150 mg; GLPG1972 75 mg; Placebo

SUMMARY:
This study is a phase 2, 52-week international, multi-regional, multi-center, randomized, double-blind, placebo-controlled dose-ranging study for the treatment of osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Male participants or female participants of non-childbearing potential and not breastfeeding.
* Body weight > 40 kg, body mass index (BMI) < 40 kg/m^2.
* Diagnosed for knee osteoarthritis based on clinical and radiological criteria of the American College of Rheumatology.
* History of knee pain for at least 6 months and on the majority of days (> 50%) during the preceding month.
* Symptom severity defined by a pain ≥ 40 mm and ≤ 90 mm on visual analogue scale (VAS, 100 mm) at screening and inclusion visits.
* Documented need for symptomatic as needed-treatment for osteoarthritis (OA) in the target knee with systemic non-steroidal anti-inflammatory drugs (NSAIDs) and/or other analgesics

Exclusion Criteria:

* Severe clinical knee malalignment according to the investigator.
* Knee prosthesis already implanted (< 1 year) or not well-tolerated (contralateral side).
* Knee prosthesis already foreseen within the study period (whichever side).
* Hip prosthesis recently implanted (< 1 year) or foreseen within the study period (whichever side).
* Previous osteotomy on the inferior limbs (whichever side).
* Surgical operation on the target knee within the 12 months prior to the screening visit or planned during the study.
* Diagnostic arthroscopy of the target knee within the 6 months prior to the screening visit or planned during the study.
* Other pathologies affecting the target knee.
* Any contraindication to magnetic resonance imaging (MRI) including the inability to undergo a knee MRI exam because of inability to fit in the scanner or knee coil.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 932 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (44):
- United States (44):
  - Central Research Associates, Inc., Birmingham, Alabama
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Hope Research Institute, LLC - Arizona, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Clinical Research Consortium Arizona, Tempe, Arizona
  - Samy Metyas MD, Inc - Covina Arthritis Clinic, Covina, California
  - TriWest Research Associates, LLC, El Cajon, California
  - BioSolutions Clinical Research Center, La Mesa, California
  - The Helm Center for Pain Management, Laguna Hills, California
  - Stanford University, Palo Alto, California
  - Artemis Institute for Clinical Research - San Diego, San Diego, California
  - Artemis Institute for Clinical Research - San Marcos, San Marcos, California
  - Encompass Clinical Research, Spring Valley, California
  - Center for Musculoskeletal Care - Yale Medicine, New Haven, Connecticut
  - Avail Clinical Research, LLC, DeLand, Florida
  - Clinical Physiology Associates Clinical Study Center, Fort Myers, Florida
  - Health Awareness, Inc, Jupiter, Florida
  - Bioclinica Research, Orlando, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Compass Research, LLC, The Villages, Florida
  - Injury Care Research, LLC, Boise, Idaho
  - Millennium Pain Center - Bloomington, Bloomington, Illinois
  - Northwestern University, Chicago, Illinois
  - Medisphere Medical Research Center, Evansville, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Phoenix Medical Reasearch, Prairie Village, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Medpharmics, Metairie, Louisiana
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Clinical Research Consortium Nevada, Las Vegas, Nevada
  - NY Scientific, Brooklyn, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Lillestol Research, LCC, Fargo, North Dakota
  - Optimed Research, LTD, Columbus, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Pioneer Research Solutions Inc., Houston, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Advanced Clinical Research, West Jordan, Utah
  - Charlottesville Medical Research Center, LCC, Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc. - Newport News, Newport News, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia

REFERENCES:
- [Derived] Chen L, Huang FL, Tang Q, Zhao ZK, Ye ZY, Liang JH. Targeted therapy for knee osteoarthritis: From basic to clinics. Medicine (Baltimore). 2025 Aug 15;104(33):e43686. doi: 10.1097/MD.0000000000043686. PMID 40826764
- [Derived] Schnitzer T, Pueyo M, Deckx H, van der Aar E, Bernard K, Hatch S, van der Stoep M, Grankov S, Phung D, Imbert O, Chimits D, Muller K, Hochberg MC, Bliddal H, Wirth W, Eckstein F, Conaghan PG. Evaluation of S201086/GLPG1972, an ADAMTS-5 inhibitor, for the treatment of knee osteoarthritis in ROCCELLA: a phase 2 randomized clinical trial. Osteoarthritis Cartilage. 2023 Jul;31(7):985-994. doi: 10.1016/j.joca.2023.04.001. Epub 2023 Apr 13. PMID 37059327
- [Derived] Brebion F, Gosmini R, Deprez P, Varin M, Peixoto C, Alvey L, Jary H, Bienvenu N, Triballeau N, Blanque R, Cottereaux C, Christophe T, Vandervoort N, Mollat P, Touitou R, Leonard P, De Ceuninck F, Botez I, Monjardet A, van der Aar E, Amantini D. Discovery of GLPG1972/S201086, a Potent, Selective, and Orally Bioavailable ADAMTS-5 Inhibitor for the Treatment of Osteoarthritis. J Med Chem. 2021 Mar 25;64(6):2937-2952. doi: 10.1021/acs.jmedchem.0c02008. Epub 2021 Mar 15. PMID 33719441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was screened on 14 August 2018. The last study visit occurred on 14 July 2020. Due to the exceptional circumstances in relation to the COVID-19 pandemic, the Sponsor decided in accordance with competent regulatory authorities' guidelines to implement some precautionary measures in order to mitigate the risk of infection.
Pre-assignment Details: A total of 3319 participants were screened and 932 participants were randomized and 931 participants were treated.
Period: Overall Study
Arm/Group | GLPG1972 75 mg | GLPG1972 150 mg | GLPG1972 300 mg | Placebo
Started | 234 | 231 | 233 | 234
Treated (All participants having taken at least one dose of investigational medicinal product (IMP)) | 234 | 231 | 232 | 234
Completed | 191 | 191 | 177 | 200
Not Completed | 43 | 40 | 56 | 34
Not completed — Adverse Event | 16 | 17 | 20 | 8
Not completed — Withdrawal by Subject | 12 | 14 | 14 | 10
Not completed — Lost to Follow-up | 6 | 4 | 5 | 6
Not completed — Protocol Violation | 2 | 0 | 6 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 2
Not completed — Miscellaneous | 7 | 5 | 10 | 6

BASELINE CHARACTERISTICS:
Population: Modified Randomised Set (mRS): All included participants to whom a therapeutic unit was randomly assigned using the interactive web response system.
Groups:
- Total: Total of all reporting groups
Arm/Group | GLPG1972 75 mg | GLPG1972 150 mg | GLPG1972 300 mg | Placebo | Total
Number analyzed (Participants) | 234 | 231 | 233 | 234 | 932
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (7.5) | 63.2 (7.2) | 62.1 (7.4) | 63.3 (7.1) | 62.9 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 165 | 154 | 163 | 646
  Male | 70 | 66 | 79 | 71 | 286
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 52 | 36 | 53 | 193
  Not Hispanic or Latino | 182 | 179 | 197 | 181 | 739
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 0 | 3
  Asian | 31 | 28 | 30 | 32 | 121
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 27 | 19 | 25 | 25 | 96
  White | 167 | 177 | 168 | 171 | 683
  More than one race | 8 | 6 | 8 | 6 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Cartilage Thickness of the Central Medial Tibiofemoral Compartment (cMTFC) of the Target Knee [Mean (Standard Deviation); unit: mm] — Cartilage thickness of the cMTFC of the target knee was measured by quantitative magnetic resonance imaging (qMRI) Population: Number of participants analyzed included participants with available data of cartilage thickness in the cMTFC at baseline.
  mm
    number analyzed (Participants) | 233 | 229 | 231 | 234 | 927
    (all) | 3.25316 (0.75857) | 3.23101 (0.75531) | 3.33075 (0.79839) | 3.18554 (0.81513) | 3.24996 (0.78289)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cartilage Thickness of the cMTFC as Assessed by qMRI on the Target Knee to Week 52
Description: Reduction in cartilage loss was assessed by cartilage thickness as measured in the medial cMTFC of the target knee using qMRI.
Time Frame: Baseline, Week 52
Population: Analysis was based on the mRS. Overall number of participants analyzed included participants with available data of cartilage thickness in the cMTFC at baseline and Week 52.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | GLPG1972 75 mg | GLPG1972 150 mg | GLPG1972 300 mg | Placebo
Number analyzed (Participants) | 162 | 158 | 151 | 172
mm | -0.06791 (0.20169) | -0.09693 (0.26839) | -0.08545 (0.21697) | -0.11562 (0.27275)
Statistical Analysis 1: Comparison: GLPG1972 75 mg vs Placebo; Estimate (Standard Error) of adjusted difference from baseline to last post baseline value between treatment groups means: GLPG1972 dose minus placebo using mixed-effects model for repeated measures (MMRM) including fixed, categorical effects of treatment, region (Asia and Rest of the World), time and treatment-by-time interaction, as well as continuous, fixed covariates of baseline and time-by-baseline interaction preceded by multiple imputation step for participants without post baseline value; Test type: Superiority; p = 0.165, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = 0.04514, 95% CI 2-sided [-0.00317 to 0.09345], Standard Error of Mean 0.02465 — Two-sided 95% confidence interval of the estimate without Dunnett adjustment
Statistical Analysis 2: Comparison: GLPG1972 150 mg vs Placebo; Estimate (Standard Error) of adjusted difference from baseline to last post baseline value between treatment groups means: GLPG1972 dose minus placebo using MMRM including fixed, categorical effects of treatment, region (Asia and Rest of the World), time and treatment-by-time interaction, as well as continuous, fixed covariates of baseline and time-by-baseline interaction preceded by multiple imputation step for participants without post baseline value; Test type: Superiority; p = 0.939, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = 0.01200, 95% CI 2-sided [-0.03868 to 0.06267], Standard Error of Mean 0.02585 — Two-sided 95% confidence interval of the estimate without Dunnett adjustment
Statistical Analysis 3: Comparison: GLPG1972 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.682, Mixed Models Analysis; Adjusted mean difference = 0.02329, 95% CI 2-sided [-0.02641 to 0.07300], Standard Error of Mean 0.02536 — Two-sided 95% confidence interval of the estimate without Dunnett adjustment

2. Secondary Outcome: Number of Participants Who Were Osteoarthritis (OA) Structural Progressors Based on Cartilage Thickness in the cMTFC Assessed by qMRI on the Target Knee
Description: A "structural progressor" was defined as a participant who had an 8% cartilage loss in cMTFC. Number of participants who met the criteria of "structural progressor" at Week 52 are provided.
Time Frame: Week 52
Population: Analysis was based on the mRS. Overall number of participants analyzed included participants with available data of cartilage thickness in the cMTFC at Week 52.
Measure: Count of Participants; unit: Participants
Arm/Group | GLPG1972 75 mg | GLPG1972 150 mg | GLPG1972 300 mg | Placebo
Number analyzed (Participants) | 162 | 158 | 151 | 172
Participants | 22 | 34 | 25 | 35
Statistical Analysis 1: Comparison: GLPG1972 75 mg vs Placebo; Estimate (Standard Error of log [estimate]) of the adjusted odds ratio between GLPG1972 dose regimen and placebo: between the proportions of participants with response: placebo versus GLPG1972 dose regimen; Test type: Superiority; p = 0.396, Logistic Model — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.84 to 2.58], Standard Error of Mean 0.29 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 2: Comparison: GLPG1972 150 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.951, Logistic Model — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.53 to 1.50], Standard Error of Mean 0.26 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 3: Comparison: GLPG1972 300 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.985, Logistic Model — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.64 to 1.83], Standard Error of Mean 0.27 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment

3. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Total Score and Subscales Scores for Pain, Function, and Stiffness to Week 52
Description: Western Ontario and McMaster Universities Osteoarthritis Index is a questionnaire designed to assess health status and health outcomes in participants with OA of the knee. The questionnaire contains 24 questions targeting areas of pain, stiffness, and physical function. Pain subscale includes 5 items rated on a Likert scale of 0 (none) to 4 (extreme) with a total range of 0-20 with higher scores indicating worse symptoms and function. Stiffness subscale includes 2 items rated on a Likert scale of 0 (none) to 4 (extreme) with a total range of 0-8 with higher scores indicating worse symptoms and function. Physical function subscale includes 17 items rated on a Likert scale of 0 (none) to 4 (extreme) with a total range of 0-68 with higher scores indicating worse symptoms and function. The total score is the sum of all subscales (range: 0 to 96) with higher scores indicating worse symptoms and function.
Time Frame: Baseline, Week 52
Population: Analysis was based on mRS. Overall number of participants analyzed included participants with available data of WOMAC score at baseline. Number of participants analyzed for change from baseline to Week 52 included participants with available data of WOMAC score at baseline and Week 52.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GLPG1972 75 mg | GLPG1972 150 mg | GLPG1972 300 mg | Placebo
Number analyzed (Participants) | 233 | 230 | 231 | 234
score on a scale
  Total score: Baseline | 48.0 (15.2) | 48.7 (15.0) | 47.0 (15.2) | 48.3 (14.5)
  Total score: Change from baseline to Week 52: number analyzed (Participants) | 189 | 187 | 176 | 200
  Total score: Change from baseline to Week 52 | -16.3 (17.7) | -16.9 (17.7) | -16.1 (19.8) | -18.4 (18.9)
  Pain subscore: Baseline | 10.2 (3.2) | 10.0 (3.1) | 9.8 (3.1) | 10.0 (3.2)
  Pain subscore: Change from baseline to Week 52: number analyzed (Participants) | 189 | 187 | 176 | 200
  Pain subscore: Change from baseline to Week 52 | -3.9 (4.1) | -3.7 (4.0) | -3.7 (4.2) | -4.1 (4.1)
  Physical function subscore: Baseline | 33.8 (11.2) | 34.3 (11.2) | 33.0 (11.6) | 34.1 (10.7)
  Physical function subscore: Change from baseline to Week 52: number analyzed (Participants) | 189 | 187 | 176 | 200
  Physical function subscore: Change from baseline to Week 52 | -11.2 (12.7) | -11.9 (13.0) | -10.9 (14.7) | -12.7 (13.9)
  Stiffness subscore: Baseline | 4.0 (1.7) | 4.3 (1.7) | 4.2 (1.6) | 4.2 (1.6)
  Stiffness subscore: Change from baseline to Week 52: number analyzed (Participants) | 189 | 187 | 176 | 200
  Stiffness subscore: Change from baseline to Week 52 | -1.2 (2.1) | -1.3 (2.0) | -1.4 (2.0) | -1.5 (2.0)
Statistical Analysis 1: Comparison: GLPG1972 75 mg vs Placebo; Total score: Estimate (Standard Error) of adjusted difference from baseline to last post baseline value between treatment groups means: placebo minus GLPG1972 dose using MMRM including fixed, categorical effects of treatment, region (Asia and Rest of the World), time and treatment-by-time interaction, as well as continuous, fixed covariates of baseline and time-by-baseline interaction preceded by multiple imputation step for participants without post baseline value; Test type: Superiority; p = 0.467, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -2.1, 95% CI 2-sided [-5.6 to 1.3], Standard Error of Mean 1.7 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 2: Comparison: GLPG1972 150 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.557, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -1.9, 95% CI 2-sided [-5.4 to 1.5], Standard Error of Mean 1.8 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 3: Comparison: GLPG1972 300 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.593, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -1.9, 95% CI 2-sided [-5.3 to 1.6], Standard Error of Mean 1.8 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 4: Comparison: GLPG1972 75 mg vs Placebo; Pain subscore: Estimate (Standard Error) of adjusted difference from baseline to last post baseline value between treatment groups means: placebo minus GLPG1972 dose using MMRM including fixed, categorical effects of treatment, region (Asia and Rest of the World), time and treatment-by-time interaction, as well as continuous, fixed covariates of baseline and time-by-baseline interaction preceded by multiple imputation step for participants without post baseline value; Test type: Superiority; p = 0.776, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -0.3, 95% CI 2-sided [-1.0 to 0.4], Standard Error of Mean 0.4 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 5: Comparison: GLPG1972 150 mg vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.446, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -0.5, 95% CI 2-sided [-1.2 to 0.3], Standard Error of Mean 0.4 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 6: Comparison: GLPG1972 300 mg vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.649, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -0.4, 95% CI 2-sided [-1.1 to 0.4], Standard Error of Mean 0.4 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 7: Comparison: GLPG1972 75 mg vs Placebo; Physical function subscore: Estimate (Standard Error) of adjusted difference from baseline to last post baseline value between treatment groups means: placebo minus GLPG1972 dose using MMRM including fixed, categorical effects of treatment, region (Asia and Rest of the World), time and treatment-by-time interaction, as well as continuous, fixed covariates of baseline and time-by-baseline interaction preceded by multiple imputation step for participants without post baseline value; Test type: Superiority; p = 0.452, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -1.6, 95% CI 2-sided [-4.1 to 0.9], Standard Error of Mean 1.3 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 8: Comparison: GLPG1972 150 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.665, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -1.2, 95% CI 2-sided [-3.7 to 1.3], Standard Error of Mean 1.3 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 9: Comparison: GLPG1972 300 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.598, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -1.3, 95% CI 2-sided [-3.9 to 1.2], Standard Error of Mean 1.3 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 10: Comparison: GLPG1972 75 mg vs Placebo; Stiffness subscore: Estimate (Standard Error) of adjusted difference from baseline to last post baseline value between treatment groups means: placebo minus GLPG1972 dose using MMRM including fixed, categorical effects of treatment, region (Asia and Rest of the World), time and treatment-by-time interaction, as well as continuous, fixed covariates of baseline and time-by-baseline interaction preceded by multiple imputation step for participants without post baseline value; Test type: Superiority; p = 0.400, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -0.2, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.2 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 11: Comparison: GLPG1972 150 mg vs Placebo; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p = 0.393, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -0.2, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.2 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 12: Comparison: GLPG1972 300 mg vs Placebo; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p = 0.858, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -0.1, 95% CI 2-sided [-0.5 to 0.2], Standard Error of Mean 0.2 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment

4. Secondary Outcome: Change From Baseline in Pain Assessment in the Target Knee as Measured by Visual Analog Scale (VAS) to Week 52
Description: The participant was asked "how would you rate the pain felt in the selected knee within the last 48 hours?". The participants rated the pain by marking the level of pain on a 100-mm VAS, with 0 being no pain and 100 being extreme pain. Higher score indicated higher pain intensity.
Time Frame: Baseline, Week 52
Population: Analysis was based on mRS. Overall number of participants analyzed included participants with available data of VAS at baseline. Number of participants analyzed for change from baseline to Week 52 included participants with available data of VAS at baseline and Week 52.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | GLPG1972 75 mg | GLPG1972 150 mg | GLPG1972 300 mg | Placebo
Number analyzed (Participants) | 234 | 231 | 233 | 234
mm
  Baseline | 63.3 (11.4) | 63.8 (11.5) | 63.3 (12.1) | 63.5 (11.0)
  Change from baseline to Week 52: number analyzed (Participants) | 191 | 185 | 178 | 199
  Change from baseline to Week 52 | -27.2 (24.3) | -25.6 (26.9) | -28.2 (27.1) | -28.9 (25.0)
Statistical Analysis 1: Comparison: GLPG1972 75 mg vs Placebo; Estimate (Standard Error) of the adjusted difference from baseline to last post baseline value between treatment groups means: placebo minus GLPG1972 dose regimen using a MMRM including the fixed, categorical effects of treatment, region (Asia and Rest of the World), time and treatment-by-time interaction, as well as the continuous, fixed covariates of baseline and time-by-baseline interaction preceded by a Multiple Imputation step for participants without post-baseline measurement; Test type: Superiority; p = 0.705, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -2.2, 95% CI 2-sided [-7.1 to 2.7], Standard Error of Mean 2.5 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 2: Comparison: GLPG1972 150 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.243, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -4.1, 95% CI 2-sided [-9.0 to 0.8], Standard Error of Mean 2.5 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 3: Comparison: GLPG1972 300 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.949, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -1.1, 95% CI 2-sided [-6.1 to 3.9], Standard Error of Mean 2.5 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment

5. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Disease Activity as Measured by VAS to Week 52
Description: The participant was asked "Considering all the ways in which your knee osteoarthritis affects you, please rate on this 100 mm scale how well you are doing today". The participants rated the disease activity by marking on a 100-mm VAS, with 0 being no pain and 100 being extreme pain. Higher score indicated higher disease activity.
Time Frame: Baseline, Week 52
Population: Analysis was based on mRS. Overall number of participants analyzed included participants with available data of PGA score at baseline. Number of participants analyzed for change from baseline to Week 52 included participants with available data of PGA score at baseline and Week 52.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | GLPG1972 75 mg | GLPG1972 150 mg | GLPG1972 300 mg | Placebo
Number analyzed (Participants) | 232 | 230 | 232 | 233
mm
  Baseline | 47.1 (18.3) | 47.9 (19.0) | 49.4 (17.5) | 50.4 (19.2)
  Change from baseline to Week 52: number analyzed (Participants) | 191 | 187 | 178 | 200
  Change from baseline to Week 52 | 19.4 (30.0) | 14.3 (30.7) | 14.1 (28.4) | 14.0 (31.3)
Statistical Analysis 1: Comparison: GLPG1972 75 mg vs Placebo; Estimate (Standard Error) of the adjusted difference from baseline to last post baseline value between treatment groups means: GLPG1972 dose regimen minus placebo using a MMRM including the fixed, categorical effects of treatment, region (Asia and Rest of the World), time and treatment-by-time interaction, as well as the continuous, fixed covariates of baseline and time-by-baseline interaction preceded by a Multiple Imputation step for participants without post-baseline measurement; Test type: Superiority; p = 0.890, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = 1.4, 95% CI 2-sided [-3.4 to 6.3], Standard Error of Mean 2.5 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 2: Comparison: GLPG1972 150 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.682, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -2.3, 95% CI 2-sided [-7.1 to 2.6], Standard Error of Mean 2.5 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 3: Comparison: GLPG1972 300 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 1.000, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = 0.1, 95% CI 2-sided [-4.8 to 5.0], Standard Error of Mean 2.5 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment

6. Secondary Outcome: Number of Participants Who Were Responders Based on the Outcome Measures in Rheumatology - Osteoarthritis Research Society International (OMERACT-OARSI) Criteria
Description: OMERACT-OARSI criteria involves improvement based on WOMAC pain and function subscales and PGA. The responders according to OMERACT-OARSI criteria were participants who had:
  * A high improvement in pain or in function ≥ 50% and absolute change ≥ 20, OR
  * Improvement in at least 2 of the 3 following:
    * Pain ≥ 20% and absolute change ≥ 10
    * Function ≥ 20% and absolute change ≥ 10
    * Patient's global assessment ≥ 20% and absolute change ≥ 10.
  WOMAC pain subscale score: range of 0 to 20, higher scores indicating more pain,
  WOMAC physical function subscale score: range of 0 to 68, higher scores indicating worse physical function),
  PGA: The participant was asked "Considering all the ways in which your knee osteoarthritis affects you, please rate on this 100 mm scale how well you are doing today". The participants rated disease activity by marking on a 100-mm VAS, with 0 being no pain and 100 being extreme pain. Higher score indicated higher disease activity.
Time Frame: Week 52
Population: Analysis was based on the mRS. Overall number of participants analyzed included participants with available data of WOMAC pain and function subscales and PGA at Week 52.
Measure: Count of Participants; unit: Participants
Arm/Group | GLPG1972 75 mg | GLPG1972 150 mg | GLPG1972 300 mg | Placebo
Number analyzed (Participants) | 189 | 187 | 176 | 200
Participants | 125 | 119 | 103 | 127
Statistical Analysis 1: Comparison: GLPG1972 75 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.991, Logistic Model — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.70 to 1.58], Standard Error of Mean 0.21 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 2: Comparison: GLPG1972 150 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.992, Logistic Model — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.64 to 1.43], Standard Error of Mean 0.21 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 3: Comparison: GLPG1972 300 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.653, Logistic Model — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.55 to 1.23], Standard Error of Mean 0.21 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment

7. Secondary Outcome: Change From Baseline in Cartilage Thickness of the Total Tibiofemoral Compartment (tTFC) of the Target Knee by qMRI to Week 52
Description: Reduction of cartilage loss was measured by cartilage thickness of the tTFC of the target knee using qMRI.
Time Frame: Baseline, Week 52
Population: Analysis was based on mRS. Overall number of participants analyzed included participants with available data of cartilage thickness of the tTFC of the target knee at baseline. Number of participants analyzed for change from baseline to Week 52 included participants with available data of cartilage thickness of the tTFC of the target knee at baseline and Week 52.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | GLPG1972 75 mg | GLPG1972 150 mg | GLPG1972 300 mg | Placebo
Number analyzed (Participants) | 232 | 229 | 231 | 234
mm
  Baseline | 6.49218 (1.02749) | 6.57424 (1.02706) | 6.51256 (0.97704) | 6.45879 (1.01774)
  Change from baseline to Week 52: number analyzed (Participants) | 162 | 158 | 150 | 172
  Change from baseline to Week 52 | -0.03572 (0.17673) | -0.02401 (0.20766) | -0.01678 (0.20934) | -0.06447 (0.23480)
Statistical Analysis 1: Comparison: GLPG1972 75 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.193, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = 0.03779, 95% CI 2-sided [-0.00448 to 0.08005], Standard Error of Mean 0.02156 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 2: Comparison: GLPG1972 150 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.256, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = 0.03580, 95% CI 2-sided [-0.00801 to 0.07962], Standard Error of Mean 0.02235 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 3: Comparison: GLPG1972 300 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.201, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = 0.03884, 95% CI 2-sided [-0.00514 to 0.08281], Standard Error of Mean 0.02243 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment

8. Secondary Outcome: Change From Baseline in Bone Area of the Medial Femoral Condyle Surface of the Target Knee by qMRI to Week 28
Time Frame: Baseline, Week 28
Population: Analysis was based on mRS. Overall number of participants analyzed included participants with available data of bone area of the medial femoral condyle surface of the target knee at baseline. Number of participants analyzed for change from baseline to Week 28 included participants with available data of bone area of the medial femoral condyle surface of the target knee at baseline and Week 28.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | GLPG1972 75 mg | GLPG1972 150 mg | GLPG1972 300 mg | Placebo
Number analyzed (Participants) | 234 | 229 | 232 | 234
mm^2
  Baseline | 2343.32026 (371.23246) | 2346.17547 (373.46086) | 2354.77368 (385.91599) | 2333.67525 (362.46041)
  Change from baseline to Week 28: number analyzed (Participants) | 202 | 191 | 190 | 210
  Change from baseline to Week 28 | 8.21893 (31.81812) | 11.11178 (33.14557) | 7.63991 (33.60899) | 11.43549 (29.60810)
Statistical Analysis 1: Comparison: GLPG1972 75 mg vs Placebo; Estimate (Standard Error) of the adjusted difference from baseline to last post baseline value between treatment groups means: Placebo minus GLPG1972 dose regimen using an analysis of covariance (ANCOVA) including the factors treatment and region with baseline as covariate and no interaction, after a Multiple Imputation for missing data; Test type: Superiority; p = 0.627, ANCOVA — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = 3.12394, 95% CI 2-sided [-3.02464 to 9.27252], Standard Error of Mean 3.13671 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 2: Comparison: GLPG1972 150 mg vs Placebo; Estimate (Standard Error) of the adjusted difference from baseline to last post baseline value between treatment groups means: Placebo minus GLPG1972 dose regimen using an ANCOVA including the factors treatment and region with baseline as covariate and no interaction, after a Multiple Imputation for missing data; Test type: Superiority; p = 0.998, ANCOVA — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = 0.46842, 95% CI 2-sided [-5.82659 to 6.76343], Standard Error of Mean 3.21111 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 3: Comparison: GLPG1972 300 mg vs Placebo; [analysis description as in outcome 8, analysis 2]; Test type: Superiority; p = 0.449, ANCOVA — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = 4.11756, 95% CI 2-sided [-2.30536 to 10.54049], Standard Error of Mean 3.27590 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment

9. Secondary Outcome: Change From Baseline in Bone Area of the Medial Femoral Condyle Surface of the Target Knee by qMRI to Week 52
Time Frame: Baseline, Week 52
Population: Analysis was based on mRS. Overall number of participants analyzed included participants with available data of bone area of the medial femoral condyle surface of the target knee at baseline. Number of participants analyzed for change from baseline to Week 52 included participants with available data of bone area of the medial femoral condyle surface of the target knee at baseline and Week 52.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | GLPG1972 75 mg | GLPG1972 150 mg | GLPG1972 300 mg | Placebo
Number analyzed (Participants) | 234 | 229 | 232 | 234
mm^2
  Baseline | 2343.32026 (371.23246) | 2346.17547 (373.46086) | 2354.77368 (385.91599) | 2333.67525 (362.46041)
  Change from baseline to Week 52: number analyzed (Participants) | 162 | 160 | 154 | 172
  Change from baseline to Week 52 | 15.45592 (31.22629) | 22.06801 (42.85848) | 20.78279 (34.96462) | 18.08990 (35.93650)
Statistical Analysis 1: Comparison: GLPG1972 75 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.789, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = 2.84781, 95% CI 2-sided [-4.51643 to 10.21205], Standard Error of Mean 3.75674 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 2: Comparison: GLPG1972 150 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.661, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -3.64759, 95% CI 2-sided [-11.19071 to 3.89553], Standard Error of Mean 3.84747 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 3: Comparison: GLPG1972 300 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.843, Mixed Models Analysis — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = -2.55176, 95% CI 2-sided [-10.04053 to 4.93701], Standard Error of Mean 3.81987 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment

10. Secondary Outcome: Change From Baseline in Joint Space Width (JSW) of the Target Knee to Week 52
Description: The JSW is the space measured between the 2 bones in the knee joint and this is assessed by x-ray.
Time Frame: Baseline, Week 52
Population: Analysis was based on mRS. Overall number of participants analyzed included participants with available data of JSW at baseline. Number of participants analyzed for change from baseline to Week 52 included participants with available data of JSW at baseline and Week 52.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | GLPG1972 75 mg | GLPG1972 150 mg | GLPG1972 300 mg | Placebo
Number analyzed (Participants) | 234 | 230 | 232 | 233
mm
  Baseline | 2.504 (0.779) | 2.500 (0.783) | 2.577 (0.840) | 2.483 (0.859)
  Change from baseline to Week 52: number analyzed (Participants) | 169 | 163 | 155 | 179
  Change from baseline to Week 52 | -0.087 (0.397) | -0.167 (0.506) | -0.113 (0.464) | -0.174 (0.470)
Statistical Analysis 1: Comparison: GLPG1972 75 mg vs Placebo; Estimate (Standard Error) of the adjusted difference from baseline to last post baseline value between treatment groups means: GLPG1972 dose regimen minus placebo using an ANCOVA including the factors treatment and region with baseline as covariate and no interaction, after a Multiple Imputation for missing data; Test type: Superiority; p = 0.141, ANCOVA — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = 0.0951, 95% CI 2-sided [-0.0028 to 0.1929], Standard Error of Mean 0.0499 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 2: Comparison: GLPG1972 150 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.981, ANCOVA — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = 0.0158, 95% CI 2-sided [-0.0861 to 0.1177], Standard Error of Mean 0.0519 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment
Statistical Analysis 3: Comparison: GLPG1972 300 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.349, ANCOVA — Two-sided adjusted p-value taking into account Dunnett adjustment (to be compared to 0.05); Adjusted mean difference = 0.0753, 95% CI 2-sided [-0.0286 to 0.1792], Standard Error of Mean 0.0529 — Two-sided 95% Confidence Interval of the estimate without Dunnett adjustment

11. Secondary Outcome: Number of Participants Who Have Used at Least 1 Systemic Analgesic During the Study
Description: Systemic analgesics included anti-inflammatory and anti-rheumatic products; analgesics; anti-diarrheals, intestinal, anti-inflammatory/anti-infective agents; and drugs for functional gastrointestinal disorders.
Time Frame: Baseline up to Week 52
Population: Analysis was based on mRS.
Measure: Count of Participants; unit: Participants
Arm/Group | GLPG1972 75 mg | GLPG1972 150 mg | GLPG1972 300 mg | Placebo
Number analyzed (Participants) | 234 | 231 | 233 | 234
Participants
  Participants with at least one treatment | 216 | 213 | 211 | 212
  Anti-inflammatory and anti-rheumatic products | 173 | 167 | 180 | 178
  Analgesics | 127 | 135 | 118 | 128
  Anti-diarrheals, intestinal anti-inflammatory/anti-infective agents | 0 | 1 | 1 | 1
  Drugs for functional gastrointestinal disorders | 1 | 0 | 0 | 0

12. Secondary Outcome: Plasma Concentrations of GLPG1972
Time Frame: Pre-dose at Weeks 4, 12, and 52; Pre-dose and one post-dose sample (2-4 hours interval) at Week 28; one post dose sample (interval 4-8 hours) at Week 40
Population: Overall number of participants included participants with available data for plasma concentrations of GLPG1972. Number of participants analyzed included participants with available data for plasma concentrations of GLPG1972 at individual timepoints. As participants in the placebo arm did not receive GLPG1972, measurement of plasma concentrations of GLPG1972 for placebo arm is not applicable.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | GLPG1972 75 mg | GLPG1972 150 mg | GLPG1972 300 mg
Number analyzed (Participants) | 217 | 210 | 194
μg/mL
  Week 4: Pre-dose | 0.445 (0.319) | 1 (0.946) | 2.013 (1.468)
  Week 12: Pre-dose: number analyzed (Participants) | 208 | 203 | 192
  Week 12: Pre-dose | 0.474 (0.685) | 0.952 (0.794) | 1.788 (1.51)
  Week 28: Pre-dose: number analyzed (Participants) | 197 | 188 | 178
  Week 28: Pre-dose | 0.457 (0.409) | 0.857 (0.696) | 1.714 (1.206)
  Week 28: 2-4 hours post-dose: number analyzed (Participants) | 199 | 188 | 182
  Week 28: 2-4 hours post-dose | 1.399 (0.668) | 2.609 (1.022) | 4.764 (1.912)
  Week 40: 4-8 hours post-dose: number analyzed (Participants) | 187 | 184 | 176
  Week 40: 4-8 hours post-dose | 1.54 (0.678) | 3.13 (1.2) | 5.664 (2.425)
  Week 52: Pre-dose: number analyzed (Participants) | 159 | 151 | 147
  Week 52: Pre-dose | 0.603 (0.6) | 1.12 (1.048) | 2.132 (1.597)

13. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Event (TEAE)
Description: TEAEs were defined as all adverse events (AEs) that occurred:
  * between first IMP intake date (included) and last visit of participant, or
  * before first IMP intake date and that worsened (in terms of intensity) or became serious according to investigator opinion between first IMP intake date (included) and last visit of participant.
  Number of participants with at least 1 TEAE (serious or non-serious) are reported.
Time Frame: Baseline up to 2-weeks after last dose of IMP (up to Week 54)
Population: Safety Set: All participants having taken at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | GLPG1972 75 mg | GLPG1972 150 mg | GLPG1972 300 mg | Placebo
Number analyzed (Participants) | 234 | 231 | 232 | 234
Participants | 174 | 177 | 174 | 174

ADVERSE EVENTS:
Time Frame: Baseline up to 2-weeks after last dose of IMP (up to Week 54)
Description: TEAEs were defined as all AEs that occurred:
  * between first IMP intake date (included) and last visit of participant, or
  * before first IMP intake date and that worsened (in terms of intensity) or became serious according to investigator opinion between first IMP intake date (included) and last visit of participant.
  Analysis was based on the safety set. All serious AEs are reported, TEAEs are reported at a threshold of 3%.
Arm/Group | GLPG1972 75 mg | GLPG1972 150 mg | GLPG1972 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/234 | 1/231 | 0/232 | 0/234
Serious Adverse Events (participants affected / at risk) | 17/234 | 17/231 | 18/232 | 18/234
Other Adverse Events (participants affected / at risk) | 114/234 | 124/231 | 105/232 | 130/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GLPG1972 75 mg (N=234) | GLPG1972 150 mg (N=231) | GLPG1972 300 mg (N=232) | Placebo (N=234)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Appendiceal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Burn infection (Infections and infestations) | 0 | 0 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Cervical cord compression (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 2
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 1
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Peritoneal cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0
Angle closure glaucoma (Eye disorders) | 0 | 0 | 0 | 1
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Depression suicidal (Psychiatric disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GLPG1972 75 mg (N=234) | GLPG1972 150 mg (N=231) | GLPG1972 300 mg (N=232) | Placebo (N=234)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 34 | 26 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 10 | 6 | 19
Nasopharyngitis (Infections and infestations) | 21 | 16 | 22 | 20
Upper respiratory tract infection (Infections and infestations) | 7 | 12 | 6 | 10
Gamma-glutamyltransferase increased (Investigations) | 3 | 2 | 16 | 4
Blood creatine phosphokinase increased (Investigations) | 12 | 7 | 9 | 8
Fall (Injury, poisoning and procedural complications) | 14 | 20 | 16 | 13
Headache (Nervous system disorders) | 15 | 12 | 11 | 9
Hypertension (Vascular disorders) | 6 | 9 | 12 | 16
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 10 | 8 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 7 | 6 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 8 | 5
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 7 | 4 | 4
Bronchitis (Infections and infestations) | 8 | 7 | 5 | 6
Urinary tract infection (Infections and infestations) | 6 | 5 | 4 | 8
Influenza (Infections and infestations) | 8 | 4 | 3 | 7
Alanine aminotransferase increased (Investigations) | 4 | 3 | 10 | 7
Aspartate aminotransferase increased (Investigations) | 4 | 2 | 10 | 6
C-reactive protein increased (Investigations) | 1 | 1 | 9 | 2
Contusion (Injury, poisoning and procedural complications) | 4 | 7 | 6 | 6
Nausea (Gastrointestinal disorders) | 3 | 7 | 11 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 7 | 4 | 7
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 7 | 4 | 7
Oedema peripheral (General disorders) | 6 | 4 | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT03595618/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT03595618/SAP_001.pdf